CLINICAL TRIAL: NCT01277445
Title: Evaluation of the Effects of Fructan Prebiotics on the Intestinal Microbiota in Humans: Human Clinical Feeding Trial.
Brief Title: Effects of Fructan Prebiotics on the Intestinal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dan Ramdath (Other Government)
Collaborators: Health Canada (Other Government); Advance Foods and Materials Network (Other); University of Ontario Institute of Technology (Other); University of Lethbridge (Other)
Responsible Party: Sponsor-Investigator, Dan Ramdath, Research Scientist, Guelph Food Research Centre
Organization: Guelph Food Research Centre (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 01B46-10-0156; NDI: 2510.10 (Other Grant/Funding Number: Agriculture and Agri-Food Canada)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Study Focus is to Define the Usual Gut Microbiota Following Prebiotic Feeding
Keywords: gut microbiome; prebiotics; immunological status; fructans
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 15g/day maltodextrin for 28 days
  Interventions: Dietary Supplement: Prebiotic
- Prebiotic (Active Comparator): Consumption of 15g/day of inulin-fructan for 28 days
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Inulin-fructan 15mg/day for 28days
  Arms: Placebo
Dietary Supplement: Prebiotic — Daily consumption of 15g inulin-fructan for 28 days

SUMMARY:
Prebiotics are carbohydrate polymers believed to improve health by stimulating beneficial gastrointestinal microbial populations. Prebiotic health claims are currently not permitted in Canada due to a lack of validating scientific data. Currently, Health Canada considers 'prebiotic' to imply a health benefit that must be substantiated. Our goal is to conduct a human clinical trial to define the impacts of fructans on the colonic microbiome as well as the physiological, psychological and immunological effects on the host.

DETAILED DESCRIPTION:
Current health claims for the fructan prebiotics focus on the bifidogenic properties of these substrates. While these claims appear to be widely accepted among nutritionists, the gut-microbiology community considers this an archaic view on these complex communities which contain in excess of 400 species of which the majority have yet to be cultivated or characterized. The bifidogenic effect associated with fructans also forms the basis of current prebiotic health claims in Canada, claims which up until now have not stood up to regulatory scrutiny The primary objective of this study is to assess the impact of frucans on the human microbiome, as well as the physiological, immunological health of the host. Information generated from this study will address both aspects of the current FOA definition of what constitutes a "prebiotic". New data generated from this study will be applicable for a new health claim for prebiotics and will provide a guide for industry demonstrating the requirements for a scientifically valid study for other submissions involving prebiotics.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 50 years
* General good health
* Participant understands the study procedures and provides informed consent (signed) to participate and authorizes the release of relevant protected health information to the study investigators

Exclusion Criteria:

* History or presence of GI disorders (Irritable bowel syndrome, colitis, Crohn's disease, colon cancer or polyps)
* Recent use of antibiotics
* Regular use of high inulin containing food products.
* Known intolerance or sensitivity to any ingredients in the study product.
* BMI >30

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota | 28 days
  various culture and non-culture methods, including molecular biology techniques will be used to determine the type and relative abundance of the gut microbione of persons fed a prebiotic compared with placebo.
Changes in Immunological Status | 28 days
  Circulating levels of cytokines associated with pro-inflammatory status and regulatory activity as well as those associated with TH1 and TH2 activity will be measured. Effects of fructans on cell population profiles in the immune system will also be determined from whole peripheral blood samples, using antibodies against B and T cells, T cell subsets, Natural Killer cells, monocytes, neutrophils and dendritic cells (DC), (including CD3, CD14, CD16, CD19, CD20, CD56)and analyzing by flow cytometry.

SECONDARY OUTCOMES:
Blood lipids | 28 days
  Blood samples will be used to assess cardiovascular disease profiles and standard biochemical biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Dan Ramdath, PhD, Study Director — Guelph Food Research Centre; Martin Kalmokoff, PhD, Study Director — Agriculture and Agri-Food Canada; Steven Traplin, MD, Study Director — Nutrasource Diagnostic Inc; Maggie Laidlaw, PhD, Principal Investigator — Nutrasource Diagnostic Inc
Locations (1):
- Nutrasoource Diagnostic Inc, Guelph, Ontario, Canada

REFERENCES:
- [Background] Gourgue-Jeannot et al. 2006. Can. J. Microbiol. 52:924-933. Brooks et al. 2009. Anaerobe 15:145-154. Costa et al. 2009 J. Microbiol. Methods 78:175-180. Lupton et al. J Nutr. 2004 134:479-82. Gibson and Roberfroid. 1995. J Nutr. 125:1401-12. Parracho et al. 2007. Proc. Nutr Soc. 66:405-11. Eckburg et al. 2005. Science 308:1635-8. Brooks et al. 2003. Can J. Microbiol. 49:589-601. Kelly et al. 2005 Trends Immunol. 26:326-33. Liu et al. 2008. Proc Natl Acad Sci U S A. 105:3951-6. Tsuji et al. 2008. Semin Immunol. 20:59-66. Reigstad et al. 2009 PLoS One 4:e5842. Jenkins et al. 2005. Metabolism 54:103-12. Jenkins et al. 1999. J. Nutr. 129:1431S-1433S. Seidel et al, 2007. Br. J. Nutr. 97:349-356. DiPenta et al. 2007. Appl.Physiol. Nutr.Metabol. 32:1025-1035. Albers et al. 2005. Br. J. Nutr. 94:452-481. Suzuki et al. 2007. Sem. Imm. 19: 127-135. Macpherson et al. 2004. Science 303: 1662-1665. Maino et al. 2004. Clinical Immunol. 110: 222- 231. Coombes and Powrie 2008. Nature Reviews Immunology 8: 435-446. Bakkerk-Zierikzee et al. 2006. Pediatr Allergy Immunol 17:134-140. Svedlund et al. 1988. Digestive Dis. & Sci. 33:129-134. Francka et al., 2005. Allergy Immunol. 136:155-158.